CLINICAL TRIAL: NCT03554018
Title: Ibuprofen With or Without Acetaminophen for Acute, Non-radicular Low Back Pain: A Randomized Trial
Brief Title: Ibuprofen With or Without Acetaminophen for Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-9182
Record Dates: First submitted 2018-05-31; First posted 2018-06-12 (Actual); Results first posted 2021-09-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Acetaminophen; Ibuprofen; Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen (Experimental): Acetaminophen 500-1000mg every 6 hours for 7 days Participants in this arm will also receive ibuprofen 600mg every 6 hours for 7 days and an educational intervention.
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen 600 mg; Behavioral: Educational intervention
- Placebo (Active Comparator): Placebo Participants in this arm will also receive ibuprofen 600mg every 6 hours for 7 days and an educational intervention.
  Interventions: Drug: Ibuprofen 600 mg; Behavioral: Educational intervention; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen 500-1000mg every 6 hours
  Arms: Acetaminophen
Drug: Ibuprofen 600 mg — Ibuprofen 600mg every 6 hours
Behavioral: Educational intervention — Research personnel will provide each patient with a 15-minute educational intervention. This will be based on NIAMS (National Institute of Arthritis and Musculoskeletal and Skin Diseases) Handout on Health: Back Pain information webpage (available at http://www.niams.nih.gov/Health_Info/Back_Pain/default.asp)
Drug: Placebo oral capsule — To match acetaminophen, patients will take one or two capsules every 6 hours
  Arms: Placebo

SUMMARY:
This is a randomized clinical trial comparing two interventions for acute low back pain:

1. Ibuprofen + acetaminophen
2. Ibuprofen + placebo

Participants will include patients who present to an emergency room for management of low back pain. Medication will be dispensed to participants at the time of emergency room discharge. Data will be collected from participants by telephone for 1 week.

ELIGIBILITY:
Inclusion Criteria:

Present to emergency room primary for management of LBP, defined as pain originating between the lower border of the scapulae and the upper gluteal folds. Flank pain, that is pain originating from tissues lateral to the paraspinal muscles, will not be included.

* Musculoskeletal etiology of low back. Patients with non-musculoskeletal etiologies such as urinary tract infection, ovarian cysts, or influenza like illness will be excluded. The primary clinical diagnosis, at the conclusion of the emergency room visit, must be a diagnosis consistent with non-traumatic, non-radicular, musculoskeletal low back pain.
* Patient is to be discharged home.
* Age 18-69
* Non-radicular pain. Patients will be excluded if the pain radiates below the gluteal folds in a radicular pattern.
* Pain duration <2 weeks (336 hours).
* Prior to the acute attack of LBP, back pain cannot occur more frequently than once per month.
* Non-traumatic LBP: no substantial and direct trauma to the back within the previous month
* Functionally impairing back pain: A baseline score of > 5 on the Roland-Morris Disability Questionnaire

Exclusion Criteria:

* Not available for follow-up
* Pregnant
* Chronic pain syndrome defined as use of any analgesic medication on a daily or near-daily basis
* Allergic to or intolerant of investigational medications

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Friedman, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibuprofen and Acetaminophen: Acetaminophen 500-1000mg every 6 hours for 7 days Participants in this arm will also receive ibuprofen 600mg every 6 hours for 7 days and an educational intervention.
  Acetaminophen: Acetaminophen 500-1000mg every 6 hours
  Ibuprofen 600 mg: Ibuprofen 600mg every 6 hours
  Educational intervention: Research personnel will provide each patient with a 15-minute educational intervention. This will be based on NIAMS (National Institute of Arthritis and Musculoskeletal and Skin Diseases) Handout on Health: Back Pain information webpage (available at http://www.niams.nih.gov/Health_Info/Back_Pain/default.asp)
- Ibuprofen and Placebo: Placebo Participants in this arm will also receive ibuprofen 600mg every 6 hours for 7 days and an educational intervention.
  Ibuprofen 600 mg: Ibuprofen 600mg every 6 hours
  Educational intervention: Research personnel will provide each patient with a 15-minute educational intervention. This will be based on NIAMS (National Institute of Arthritis and Musculoskeletal and Skin Diseases) Handout on Health: Back Pain information webpage (available at http://www.niams.nih.gov/Health_Info/Back_Pain/default.asp)
  Placebo oral capsule: To match acetaminophen, patients will take one or two capsules every 6 hours
Period: Overall Study
Arm/Group | Ibuprofen and Acetaminophen | Ibuprofen and Placebo
Started | 60 | 60
Completed | 57 | 53
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen and Acetaminophen | Ibuprofen and Placebo | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (12) | 41 (13) | 41 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 31 | 32 | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120
Duration of low back pain [Median (Inter-Quartile Range); unit: hours] | 48 [24 to 96] | 48 [12 to 96] | 48 [24 to 96]

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Impairment as Measured by the Roland Morris Disability Questionnaire
Description: The Roland Morris Disability Questionnaire (RMDQ) is a 24 item instrument that evaluates the impact of low back pain on one's daily life. It is most sensitive for patients with mild to moderate disability due to acute, sub-acute or chronic low back pain. Each question can be answered as either a "yes" or "no". The score ranges from 0 to 24 where a higher score reflects greater impairment and, therefore, worsening in the quality of life. The change in RMDQ is obtained by subtracting the RMDQ score at one week after discharge from the baseline score. The calculated mean and associated confidence interval values have been verified by staff statisticians.
Time Frame: Baseline and one week after discharge from emergency department
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibuprofen and Acetaminophen | Ibuprofen and Placebo
Number analyzed (Participants) | 57 | 53
units on a scale | 11.1 (10.7) | 11.9 (9.7)

2. Secondary Outcome: Number of Participants With Moderate or Severe Pain, as Measured on an Ordinal Scale
Description: Data collected by telephone questionnaire. Participants asked to assess intensity of low back pain over the previous 24 hours, using a four point ordinal scale: severe, moderate, mild, or none.
Time Frame: 7 days after discharge from emergency department
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen and Acetaminophen | Ibuprofen and Placebo
Number analyzed (Participants) | 57 | 53
Participants | 16 | 15

3. Secondary Outcome: Number of Participants Who Required Analgesic Medication for Low Back Pain Within the Previous 24 Hours.
Description: Telephone questionnaire is used to assess number of patients needing any analgesic or low back pain medication within the previous 24 hours.
Time Frame: 7 days after discharge from emergency department
Population: Data was collected and analyzed for 52 participants in the "Ibuprofen and Placebo" group.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen and Acetaminophen | Ibuprofen and Placebo
Number analyzed (Participants) | 57 | 52
Participants | 36 | 32

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Ibuprofen and Acetaminophen | Ibuprofen and Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 5/60 | 2/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibuprofen and Acetaminophen (N=60) | Ibuprofen and Placebo (N=60)
Diarrhea (Gastrointestinal disorders) | 3 | 1
Drowsiness (Nervous system disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT03554018/Prot_SAP_000.pdf